CLINICAL TRIAL: NCT04208763
Title: Imipenem and Tigecycline Versus Imipenem and Tigecycline With GM-CSF for the Management of Spontaneous Bacterial Peritonitis Presenting With Septic Shock.
Brief Title: A Randomized Controlled Trial Comparing Imipenem and Tigecycline Versus Imipenem and Tigecycline With GM-CSF for the Management of Spontaneous Bacterial Peritonitis Presenting With Septic Shock.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-SBP-02
Record Dates: First submitted 2019-12-12; First posted 2019-12-23 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Imipenem; Tigecycline; Colistin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imipenem+Tigecycline+GM-CSF (Experimental)
  Interventions: Drug: Imipenem; Drug: Tigecycline; Drug: GMCSF; Drug: Colistin
- Imipenem+Tigecycline (Active Comparator)
  Interventions: Drug: Imipenem; Drug: Tigecycline; Drug: Colistin

INTERVENTIONS:
Drug: Imipenem — Inj Imipenem 1gm i.v. TDS
Drug: Tigecycline — Inj Tigecycline 100mg stat f/b 50mg i.v. OD
Drug: GMCSF — Inj GM-CSF 500mcg s.c. OD
  Arms: Imipenem+Tigecycline+GM-CSF
Drug: Colistin — Inj Colistin 9 MIU i.v. stat f/b 4.5 MIU i.v. BD

SUMMARY:
Study population: A total of 90 consecutive patients of decompensated cirrhosis of any etiology, presenting to the Institute of Liver and Biliary Sciences with SBP with septic shock will be included.

Study design: Randomized controlled trial Study period: August 2019 to December 2021. Sample size: Assuming that the response rate is 90% with GM-CSF and 60% without GM-CSF after day 5. With alpha 5 and power 80,we need to enroll 76 cases (38 cases with each). Further assuming 20 % drop-out due to various reasons, it was decided to enroll 90 cases randomly allocated into two groups (i.e., 45 in each) by block randomization method by taking block size as 6. So for the present study, it was decided to enroll 90 cases in all.

Group A will be given Imipenem and Tigecycline. Patients with recent hospitalisation will be given Colistin in addition.

Group B will be given: To another group we will give Imipenem and Tigecycline and GMCSF.Patients with recent hospitalisation will be given Colistin in addition.

The dose of antibiotic will be given at dosage Inj Imipenem 1gm i.v. TDS Inj Tigecycline 100mg stat f/b 50mg i.v. OD Inj GM-CSF 500mcg s.c. OD Inj Colistin 9 MIU i.v. stat f/b 4.5 MIU i.v. BD Monitoring and assessment At the baseline, all patients will undergo investigational evaluation as described

Daily monitoring of following parameters:

* Haemoglobin,
* Total peripheral leucocyte counts,
* Platelet counts,
* Renal function tests
* Liver function tests and
* Chest X rays will be undertaken
* Ascitic fluid analysis will be done on day 0, day 2 and day 5

Stopping rule:If the patient develops a TLC of more than 50,000, the dose of the GM CSF will be reduced to half and the treatment continued. If, even after the reduction, the TLC rises to more than 50,000, then the treatment will be stopped and the patient excluded.

Expected outcome of the project: Addition of GM-CSF to standard antibiotic regimen helps resolve SBP and improves outcome in decompensated liver cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Spontaneous Bacterial Peritonitis (SBP) with shock in a cirrhotic
2. Hospital acquired SBP with shock
3. Difficult to treat SBP

Exclusion Criteria:

1. Refractory Shock
2. Cardiac comorbidities (known Coronary Artery Disease)
3. Chronic Kidney Disease on Maintenance Hemodialysis
4. < 18 years.
5. Advanced Hepatocellular Carcinoma
6. Post liver transplant
7. HIV + ve, Immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of Spontaneous Bacterial peritonitis in both groups | Day 5
  Response is defined by resolution of SBP in terms of total counts < 500,Neutrophil<250

SECONDARY OUTCOMES:
Reversal of shock in both groups | Day 2
  Blood pressure more than 90/60 mmHg with no inotropes requirement
Survival in both groups | Day 7
Survival in both groups | Day 28
Change in ascitic fluid metabolites Nitric Oxide in both groups | Day 28
  change is defined as percentage reduction in nitric oxide
Change in ascitic fluid macrophage population in both groups | Day 28
  change is defined as percentage reduction in macrophage population
Development of Hepatic Encephalopathy in both groups. | Day 28
  Hepatic Encephalopathy will be measured as per West Haven criteria
Development of Acute Kidney Injury in both groups | Day 28
  AKIN criteria will be used for Acute kidney injury
Development of Pneumonia in both groups. | Day 28
  Pneumonia will be confirmed based on imaging and clinically
Development of organ failures in both groups. | Day 28
  Organ failure will be as per APACHE score
Development of coagulopathy in both groups. | Day 28
  Coagulopathy is defined as INR > 1.5
Resolution of Spontaneous Bacterial peritonitis in both groups | Day 2
  Response is defined by resolution of SBP in terms of total counts < 500,Neutrophil<250

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided